CLINICAL TRIAL: NCT04528212
Title: Comparison of the Effect of Fenofibrate Versus Curcumin in Type 2 Diabetic Patients Treated With Glimepiride
Brief Title: Fenofibrate Versus Curcumin in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Principal Investigator, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fenofibrate vs curcumin
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Fenofibrate; Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Glimepiride (4 mg) per Day
  Interventions: Drug: Glimepiride Tablets
- Group II (Experimental): Glimepiride (4 mg) plus Fenofibrate (160 mg) per Day
  Interventions: Drug: glimepiride plus fenofibrate
- Group III (Experimental): Glimepiride (4 mg) plus Curcumin (1100 mg) With 5mg Black Pepper per Day
  Interventions: Drug: glimepiride plus curcumin

INTERVENTIONS:
Drug: Glimepiride Tablets — Glimepiride (4 mg) per Day
  Other Names: Amaryl 4 mg
  Arms: Group I
Drug: glimepiride plus fenofibrate — Glimepiride (4 mg) plus Fenofibrate (160 mg) per Day
  Other Names: Amaryl 4 mg Plus Lipanthyl Supra (160 mg)
  Arms: Group II
Drug: glimepiride plus curcumin — Glimepiride (4 mg) plus Curcumin (1100 mg) With 5mg Black Pepper per Day
  Other Names: Amaryl 4 mg Plus Curcumin (1100 mg) With 5mg Black Pepper
  Arms: Group III

SUMMARY:
The aim of this study is to evaluate the effect of fenofibrate versus curcumin on glycemic status, lipids profile, hs-CRP, sirtuin-1 and fetuin-A in type 2 diabetic patients who are taking glimepiride.

DETAILED DESCRIPTION:
Method & Proposal Steps

1- Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University. 2- All participants agreed to take part in this clinical study and provide informed consent. 3- (60) Patients with DM type 2 who's taking Glimepiride will be enrolled from Internal Medicine Department, Tanta University Hospital. 4- Serum samples will be collected for measuring the biomarkers. 5- All enrolled patients will be mentioned as two groups; Group I are patients who will be prescribed glimepiride plus fenofibrate. Group II are patients who will be prescribed glimepiride plus curcumin. 6- All patients will be followed up during 3 months' period. 7- At the end of 3 months on the new regimen, steps 4 will be repeated. 8- Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results. 9- Measuring outcome: The primary outcome is the change of serum levels of the measured markers after 3 months and lipid profile. 10- Results, conclusion, discussion and recommendations will be given.

Methodology Serum levels of fetuin-A, and Sirtuin1 (SIRT1) will be measured ELISA. Lipid profile. Fasting Blood glucose and 2 hrs postprandial Blood Glucose. Hb A1C will be measured. BMI of the patients will be measured before and after the study. High sensitivity C-reactive protein (hs-CRP) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 60 Patients with type 2 DM diagnosed clinically.
* The age ranged from 35 to 70 years.
* There are no limits to the duration of DM and gender.
* HbA1c ≥ 7

Exclusion Criteria:

1. Other types of DM
2. Hypersensitivity to the drug
3. Abnormal liver function
4. Patients with renal impairment (eGFR ≤ 60 ml/min)
5. Addition of any antidiabetic medications or insulin during follows up.
6. Pregnancy, lactation or child-bearing potential. 7. No insulin therapy and no use of antioxidants, multivitamin.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
fetuin-A (mg/L) | three months
  human Fetuin A protein
Sirtuin1 (SIRT1) (ng/ml) | three months
  human Sirtuin1 a Protein - Recombinant human SIRT1 protein

SECONDARY OUTCOMES:
Total Cholesterol (mg/dl) | Three Months
  Total Cholesterol
Triglyceride (mg/dl) | Three Months
  Triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass.Prof., Study Chair — Damanhour University; Eman Nada, B. Pharm, Principal Investigator — Damanhour University; Haidy Abass, Ass.Prof., Study Director — Damanhour University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Panahi Y, Khalili N, Sahebi E, Namazi S, Reiner Z, Majeed M, Sahebkar A. Curcuminoids modify lipid profile in type 2 diabetes mellitus: A randomized controlled trial. Complement Ther Med. 2017 Aug;33:1-5. doi: 10.1016/j.ctim.2017.05.006. Epub 2017 May 29. PMID 28735818
- [Result] Poolsup N, Suksomboon N, Kurnianta PDM, Deawjaroen K. Effects of curcumin on glycemic control and lipid profile in prediabetes and type 2 diabetes mellitus: A systematic review and meta-analysis. PLoS One. 2019 Apr 23;14(4):e0215840. doi: 10.1371/journal.pone.0215840. eCollection 2019. PMID 31013312 (Retraction: PMID 32442218 PLoS One. 2020 May 22;15(5):e0233919)
- [Result] Noureldein MH, Abd El-Razek RS, El-Hefnawy MH, El-Mesallamy HO. Fenofibrate reduces inflammation in obese patients with or without type 2 diabetes mellitus via sirtuin 1/fetuin A axis. Diabetes Res Clin Pract. 2015 Sep;109(3):513-20. doi: 10.1016/j.diabres.2015.05.043. Epub 2015 Jun 11. PMID 26105582
- [Derived] Nada EM, El-Gharbawy NM, Abbas H, Werida RH. Effect of adding fenofibrate versus curcumin to glimepiride in patients with type 2 diabetes: a randomized controlled trial. BMC Pharmacol Toxicol. 2025 Jun 6;26(1):119. doi: 10.1186/s40360-025-00950-y. PMID 40481568